CLINICAL TRIAL: NCT05267132
Title: Adolescent Acts of Kindness Intervention With Reflection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Andrew J. Fuligni, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB#21-002091
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Wellness 1
Keywords: adolescence; psychological well-being; social connection; kindness
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: 120 participants will randomly be assigned to one of three conditions. Participants will complete a 4-week intervention. All outcomes will be measured before and after the intervention, and some psychological measures will be collected weekly throughout the intervention.
Who Masked: Participant
Masking Description: Participants will be told that the investigators are studying the daily lives of teens. They will not be informed of the other arms of the experiment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Kindness to Others with Reflection (Experimental): Participants will complete the 'Other-Focused Acts of Kindness Intervention' by performing acts of kindness for others and will also complete a reflection component. They will be asked to complete 3 kind acts for others throughout the week for 4 weeks. They will receive text messages three days per week (either Tuesday, Thursday, and Saturday or Wednesday, Friday, and Sunday) and will report on their kind act later that day. At the end of each intervention week, they will be asked to reflect upon their experience of performing kind acts for others.
  Interventions: Behavioral: Other-Focused Acts of Kindness Intervention with Reflection
- Kindness to Others (Active Comparator): Participants will complete the 'Other-Focused Acts of Kindness Intervention' by performing acts of kindness for others. They will be asked to complete 3 kind acts for others throughout the week for 4 weeks. They will receive text messages three days per week (either Tuesday, Thursday, and Saturday or Wednesday, Friday, and Sunday) and will report on their kind act later that day.
  Interventions: Behavioral: Other-Focused Acts of Kindness Intervention
- Daily Report (Sham Comparator): Participants will complete the 'Daily Reports' and be asked to report their daily activities throughout the week for 4 weeks. They will receive text messages three days per week (either Tuesday, Thursday, and Saturday or Wednesday, Friday, and Sunday) and will list activities from their day.
  Interventions: Behavioral: Daily Reports

INTERVENTIONS:
Behavioral: Other-Focused Acts of Kindness Intervention with Reflection — Participants engage in positive behaviors by completing acts of kindness for others three times per week. These acts should require effort and be outside of an individual's normal routine. Participants will then reflect on their kind acts after each week.
  Arms: Kindness to Others with Reflection
Behavioral: Other-Focused Acts of Kindness Intervention — Participants engage in positive behaviors by completing acts of kindness for others three times per week. These acts should require effort and be outside of an individual's normal routine.
  Arms: Kindness to Others
Behavioral: Daily Reports — Participants will report their daily activities three times per week. Aside from reporting at the end of the day, no changes should be made to the individual's normal routine.
  Arms: Daily Report

SUMMARY:
Adolescents will complete a 4-week intervention, during which they will either complete a kind act for others, complete a kind act for others with a reflection component, or report their daily activities three days per week. Psychological measures will be indexed before and after the intervention.

DETAILED DESCRIPTION:
There is growing policy and scientific interest in promoting the positive benefits of kindness and prosociality. This is particularly true for adolescents, whose psychological and social maturation offers fertile ground in which kindness can be seeded early in life with potentially positive effects on their psychological health. Much of the existing efforts have focused on large-scale community engagement and service-learning programs. Investigating less costly and time-intensive alternatives is necessary to broaden engagement and access. This project aims to implement one such effort with an enhanced acts of kindness intervention for adolescents. The enhancement incorporates existing evidence that requiring adolescents to reflect upon and savor their experience of helping others promotes the positive impact of such interventions. 120 high-school-aged youth will be recruited and assigned to one of three groups (40/group). Participants will either conduct a kind act for others, complete a kind act for others with a reflection component (enhanced condition), or report their daily activities three days per week for 4 weeks. During this intervention, they will receive text messages 3 days per week instructing them to complete their respective act. Participants will provide a brief description of this act that evening, as well as complete brief surveys at the end of the week for each week of the intervention. Participants will also complete a pre- and post-intervention questionnaire and participants' parents will complete a brief survey at the start of the study to provide demographic information and an idea of what prosocial behaviors participants witnessed in their home. The investigators will use these data to assess the effects of prosocial behavior on psychological health. Conceptual frameworks from developmental psychology guide the hypothesis that prosocial behavior will influence adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 14-17

Exclusion Criteria:

* None

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Average Positive Affect | Weekly over 5 weeks
  Average Positive Affect as assessed by the positive affect subscale of the Affect Adjective Checklist. An average is taken across four items, and scores range from 1 to 5 with higher scores indicating more positive affect over the week.

SECONDARY OUTCOMES:
Average Psychological Flourishing | Baseline and one-week post intervention (elapsed time of 5 weeks)
  Change in average psychological flourishing from baseline to one week following the intervention as assessed by Mental Health Continuum-Short Form at week 5. An average is taken across 20 items, and scores range from 1 to 6, with higher values representing greater psychological flourishing.
Average Negative Affect | Weekly over 5 weeks
  Average negative affect as assessed by the negative affect subscale of the Affect Adjective Checklist. An average is taken across five items, and scores range from 1 to 5 with higher scores indicating more negative affect over the week.

OTHER OUTCOMES:
Average Stress | Weekly over 5 weeks
  Average stress as assessed by the Perceived Stress Scale. An average is taken across 10 items, and scores range from 1 to 5 with higher scores indicating greater stress.
Sleep Quality | Weekly over 5 weeks
  Sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI). The assessment has 7 components, each scored from 0 to 3. A sum is taken across these components, such that total scores range from 0 to 21 with higher scores indicating poorer sleep.
Average Social Connection | Weekly over 5 weeks
  Average social connection as assessed by the relatedness subscale of the Balanced Measure of Psychological Needs. An average is taken across 6 items, and scores range from 1 to 5 with higher scores indicating greater social connection.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Fuligni, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Adolescent Development Lab, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No